CLINICAL TRIAL: NCT02590718
Title: Management Following Lumbar Puncture In Children
Acronym: MFLPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Gang Liu, Chief physician/Professor, Beijing Children's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20150826
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Spinal Puncture Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): optimized postoperative management(lying without the pillow for half an hour after lumbar puncture)
  Interventions: Procedure: optimized postoperative management
- Group 2 (No Intervention): traditional postoperative management(lying without the pillow and fasting water and food for four hours after lumbar puncture)

INTERVENTIONS:
Procedure: optimized postoperative management — lying without the pillow for half an hour after lumbar puncture
  Arms: Group 1

SUMMARY:
The study is carried out in a prospectively randomly controlled way. In the context of acknowledgement and understanding from parents, by comparing with traditional process (lying without the pillow and fasting water and food for four hours following lumbar puncture), an optimized postoperative management (lying without the pillow for half an hour following lumbar puncture) is randomly selected. All children will be evaluated by the FLACC (The face, legs, activity, cry, consolability behavioral tool) scale to assess the degree of pain after lumbar puncture. Any postoperative condition will be recorded and analyzed. A questionaire about bad memory during lumbar puncture for all parents and children will be investigated in order to establish an optimized lumbar puncture management process.

DETAILED DESCRIPTION:
The purpose of this study is to establish an optimized lumbar puncture management process on the basis of fully understanding of parents and children. An improved process consisting of comfortable LP will be established upon completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* children with indications of lumbar puncture;
* voluntarily signed the informed consent

Exclusion Criteria:

* topical anesthetic skin allergies;
* skin infection in lumbar puncture site;
* severe intracranial hypertension;
* unstable vital signs;
* coagulopathy;
* intracranial hemorrhage and occupying;
* low back pain;
* headache and low back pain before lumbar puncture;
* past headache after lumbar puncture;
* mental retardation, neuropsychiatric symptoms;
* children could not immediately act after the lumbar puncture(such as disturbance of consciousness or suffering from underlying diseases or drainage);
* the case with repeated puncture in one operation

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Postoperation complications include headache, backache, vomit, cerebral hernia etc. | up to five days postoperation

SECONDARY OUTCOMES:
Composite measure of Vital signs include heart rate, pulse, blood pressure and respiration. | up to four hours postoperation
comfort degree | up to four hours postoperation
  evaluated by the FLACC(The face,legs,activity,cry,consolability behavioral tool) scale
whether bad memories exist or not | up to four hours postoperation
  A questionaire about the operation for all parents and children will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Liu, MD, Principal Investigator — Beijing Childrens' Hospital

REFERENCES:
- [Derived] Hu B, Chen TM, Liu B, Chi W, Miao YQ, Nie XL, Peng XX, Liu G. Optimal management after paediatric lumbar puncture: a randomized controlled trial. BMC Neurol. 2019 Apr 13;19(1):64. doi: 10.1186/s12883-019-1275-9. PMID 30987603